CLINICAL TRIAL: NCT03340571
Title: mtDNA Damage in Alzheimer's Disease (AD)
Brief Title: Blood Biomarker of Alzheimer's Disease (AD)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00085997
Record Dates: First submitted 2017-11-09; First posted 2017-11-13 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; biomarkers; blood
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Alzheimer's Patients
- Healthy Volunteers

SUMMARY:
Currently, no cures or disease modifying therapies exist for Alzheimer's disease (AD). This is partially due to the inability to detect the disease before it has progressed to a stage where there are clinical manifestations. The identification and validation of high throughput biomarkers to measure disease progression (as well as identify pre-clinical disease onset) is critical to the development of disease-modifying or even preventative therapies. In this study, we are testing a blood biomarker for stratification of Alzheimer's disease patients and healthy volunteers. This study may lead to future blood tests that may help earlier diagnosis of Alzheimer's disease and detect the disease progression.

ELIGIBILITY:
Inclusion Criteria:

Alzheimer's Disease Patients:

* 50 years and older
* AD patient who is seen at the Memory Disorders Clinic
* AD diagnosis
* Non smoking
* No cancer treatment in the last 5 years
* Informed consent from the patient or the patient's legally authorized representative (LAR)
* Patient and/or LAR able to read and speak English

Healthy Control Participants:

* 50 years and older
* Non smoking
* No cancer treatment in the last 5 years
* Age matched to AD subject
* Able to read and speak English

Exclusion Criteria:

Alzheimer's Disease Patients:

* Known additional neurological disease

Healthy Control Participants:

* Neurological degenerative diseases (such as Parkinson's, Alzheimer's or Huntington's)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research coordinator(s) will review the clinic schedule in the Memory Disorders clinic at Duke University for potential patients who meet the basic inclusion/exclusion criteria who have appointments that day.
  While consenting AD potential subjects, the study team may also ask their caregivers who accompany the AD patient to the clinic if they would also like to be part of the study and possibly enroll as a Healthy Control subject.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Biological marker of Alzheimer's disease | Day 1
  Test for blood biological marker of Alzheimer's disease, mtDNA damage

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Sanders, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No